CLINICAL TRIAL: NCT00396539
Title: Detection of Hydrogen Sulfide Production by Oral Microflora Samples
Brief Title: Hydrogen Sulfide Production by Oral Microflora
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 29.12.06-19-HMO-CTIL
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2006-11

CONDITIONS: Oral Malodor (Halitosis)
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Oral malodor is a common condition. In most cases this condition results from the proteolytic activity of anaerobic oral bacteria. These bacteria produce volatile sulfide compounds which are fowl smelling and are felt during exhalation and speech. the aim of the present study is to examine a simple method of detecting these bacteria in samples taken from the oral cavity of oral malodor patients.

ELIGIBILITY:
Inclusion Criteria:

* oral malodor patients

Exclusion Criteria:

* smokers, users of antibiotic one month prior to study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nir Sterer, Dr., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel